CLINICAL TRIAL: NCT04462315
Title: Ten-year Follow-up of the Clinical Evaluation of Everolimus-Eluting Coronary Stents in the Treatment of Patients With ST-segment Elevation Myocardial Infarction: EXAMINATION-EXTEND Trial
Brief Title: 10-Years Follow-up of the EXAMINATION Trial
Acronym: EXAMINAT10N
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: HCB/2018/0906
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2020-07

CONDITIONS: Myocardial Infarction; ST Elevation Myocardial Infarction; Infarction; Necrosis; Heart Disease; Cardiovascular Diseases; Vascular Diseases
Keywords: Acute myocardial infarction; Primary Percutaneous Coronary Intervention; Drug-Eluting Stent
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Infarction; Necrosis; Heart Diseases; Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Everolimus Arm: Everolimus Eluting Coronary Stent System
  Interventions: Drug: Everolimus Eluting Coronary Stent System
- Non-drug eluting stent Arm: Cobalt chromium balloon-expandable stent
  Interventions: Device: Cobalt chromium balloon expandable stent (non-drug-eluting stent Arm)

INTERVENTIONS:
Drug: Everolimus Eluting Coronary Stent System — Everolimus Eluting Coronary Stent System (Everolimus Arm) implantation
  Other Names: N/H
  Groups: Everolimus Arm
Device: Cobalt chromium balloon expandable stent (non-drug-eluting stent Arm) — Cobalt chromium balloon-expandable stent (non-drug-eluting stent Arm) implantation
  Other Names: N/H
  Groups: Non-drug eluting stent Arm

SUMMARY:
The EXAMINATION trial was a superiority trial that compared everolimus-eluting stents (EES) versus bare-metal stents (BMS) in an all-comer ST-segment elevation myocardial infarction (STEMI) population. The patient-oriented endpoint was not superior at 1-year, but it was at 5-year. However, very-long term follow-up is unknown. The study had an independent Clinical event Committee (CEC). All events were adjudicated by an independent clinical committee, according to the Academic Research Consortium 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were enrolled in the EXAMINATION trial (NCT00828087).

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The EXAMINATION trial population was an all-comers population with ST-elevation myocardial infarction, representative of routine clinical practice.
Sampling Method: Probability Sample
Enrollment: 1498 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Patient-oriented Composite Endpoint (PoCE) | 10 years
  Rate of composite endpoint of all-cause death, any myocardial infarction, and any revascularization. Defined according to the Academic Research Consortium 1.

SECONDARY OUTCOMES:
Device-oriented Composite Endpoint (DoCE) | 10 years
  Rate of composite endpoint of cardiac death, Target vessel myocardial infarction, and Target lesion revascularization. Defined according to the Academic Research Consortium 1.
Rate of all cause and cardiac mortality | 10 years
  Defined according to the Academic Research Consortium 1.
Rate of recurrent myocardial infarction | 10 years
  Defined according to the Academic Research Consortium 1.
Rate of target lesion revascularization | 10 years
  Defined according to the Academic Research Consortium 1.
Rate of stent thrombosis | 10 years
  Defined according to the Academic Research Consortium 1.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Brugaletta, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona; Josep Gómez-Lara, MD, PhD, Principal Investigator — Hospital Universitari de Bellvitge; Luis Ortega-Paz, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona; Manel Sabaté, MD, PhD, Study Chair — Hospital Clinic of Barcelona
Locations (11):
- Italy (2):
  - Azienda Ospedaliera Bolognini, Seriate, Bergamo
  - Azienda Ospedaliero Universitaria S. Anna di Ferrara, Ferrara
- Erasmus MC, Rotterdam, Rotterdam, Netherlands
- Spain (8):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Clínic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital de Bellvitge, Barcelona, Catalonia
  - Complejo Hospitalario U. A Coruña, A Coruña, Galicia
  - Hospital Álvaro Cunqueiro, Vigo, Galicia
  - Hospital Son Dureta, Palma de Mallorca, Mallorca
  - Hospital General de Alicante, Alicante, Valencia
  - Hospital Clínico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No
Will be made available upon request.

REFERENCES:
- [Background] Sabate M, Cequier A, Iniguez A, Serra A, Hernandez-Antolin R, Mainar V, Valgimigli M, Tespili M, den Heijer P, Bethencourt A, Vazquez N, Brugaletta S, Backx B, Serruys P. Rationale and design of the EXAMINATION trial: a randomised comparison between everolimus-eluting stents and cobalt-chromium bare-metal stents in ST-elevation myocardial infarction. EuroIntervention. 2011 Dec;7(8):977-84. doi: 10.4244/EIJV7I8A154. PMID 22115622
- [Background] Sabate M, Cequier A, Iniguez A, Serra A, Hernandez-Antolin R, Mainar V, Valgimigli M, Tespili M, den Heijer P, Bethencourt A, Vazquez N, Gomez-Hospital JA, Baz JA, Martin-Yuste V, van Geuns RJ, Alfonso F, Bordes P, Tebaldi M, Masotti M, Silvestro A, Backx B, Brugaletta S, van Es GA, Serruys PW. Everolimus-eluting stent versus bare-metal stent in ST-segment elevation myocardial infarction (EXAMINATION): 1 year results of a randomised controlled trial. Lancet. 2012 Oct 27;380(9852):1482-90. doi: 10.1016/S0140-6736(12)61223-9. Epub 2012 Sep 3. PMID 22951305
- [Background] Sabate M, Brugaletta S, Cequier A, Iniguez A, Serra A, Jimenez-Quevedo P, Mainar V, Campo G, Tespili M, den Heijer P, Bethencourt A, Vazquez N, van Es GA, Backx B, Valgimigli M, Serruys PW. Clinical outcomes in patients with ST-segment elevation myocardial infarction treated with everolimus-eluting stents versus bare-metal stents (EXAMINATION): 5-year results of a randomised trial. Lancet. 2016 Jan 23;387(10016):357-366. doi: 10.1016/S0140-6736(15)00548-6. Epub 2015 Oct 29. PMID 26520230
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Derived] Verardi FM, Bujak K, Tolomeo P, Gomez-Lara J, Jimenez-Diaz V, Jimenez M, Jimenez-Quevedo P, Diletti R, Bordes P, Campo G, Silvestro A, Maristany J, Flores X, de Miguel-Castro A, Iniguez A, Ielasi A, Tespili M, Lenzen M, Gonzalo N, Tebaldi M, Biscaglia S, Vidal-Cales P, Ortega-Paz L, Romaguera R, Gomez-Hospital JA, Serruys PW, Sabate M, Brugaletta S. Ten-year prognostic impact of target versus non-target vessel failure after STEMI. Insight from the EXAMINATION-EXTEND trial. Rev Esp Cardiol (Engl Ed). 2024 Mar;77(3):215-225. doi: 10.1016/j.rec.2023.07.001. Epub 2023 Jul 26. English, Spanish. PMID 37506972
- [Derived] Spione F, Arevalos V, Gabani R, Ortega-Paz L, Gomez-Lara J, Jimenez-Diaz V, Jimenez M, Jimenez-Quevedo P, Diletti R, Pineda J, Campo G, Silvestro A, Maristany J, Flores X, Oyarzabal L, Bastos-Fernandez G, Iniguez A, Serra A, Escaned J, Ielasi A, Tespili M, Lenzen M, Gonzalo N, Bordes P, Tebaldi M, Biscaglia S, Al-Shaibani S, Romaguera R, Gomez-Hospital JA, Rodes-Cabau J, Serruys PW, Sabate M, Brugaletta S. Impact of Diabetes on 10-Year Outcomes Following ST-Segment-Elevation Myocardial Infarction: Insights From the EXAMINATION-EXTEND Trial. J Am Heart Assoc. 2022 Dec 6;11(23):e025885. doi: 10.1161/JAHA.122.025885. Epub 2022 Nov 29. PMID 36444863
- [Derived] Gabani R, Spione F, Arevalos V, Grima Sopesens N, Ortega-Paz L, Gomez-Lara J, Jimenez-Diaz V, Jimenez M, Jimenez-Quevedo P, Diletti R, Pineda J, Campo G, Silvestro A, Maristany J, Flores X, Oyarzabal L, Bastos-Fernandez G, Iniguez A, Serra A, Escaned J, Ielasi A, Tespili M, Lenzen M, Gonzalo N, Bordes P, Tebaldi M, Biscaglia S, Al-Shaibani S, Romaguera R, Gomez-Hospital JA, Rodes-Cabau J, Serruys PW, Sabate M, Brugaletta S. Sex Differences in 10-Year Outcomes Following STEMI: A Subanalysis From the EXAMINATION-EXTEND Trial. JACC Cardiovasc Interv. 2022 Oct 10;15(19):1965-1973. doi: 10.1016/j.jcin.2022.07.038. Epub 2022 Aug 22. PMID 36008267
- [Derived] Brugaletta S, Gomez-Lara J, Ortega-Paz L, Jimenez-Diaz V, Jimenez M, Jimenez-Quevedo P, Diletti R, Mainar V, Campo G, Silvestro A, Maristany J, Flores X, Oyarzabal L, De Miguel-Castro A, Iniguez A, Serra A, Nombela-Franco L, Ielasi A, Tespili M, Lenzen M, Gonzalo N, Bordes P, Tebaldi M, Biscaglia S, Rodriguez-Arias JJ, Al-Shaibani S, Arevalos V, Romaguera R, Gomez-Hospital JA, Serruys PW, Sabate M. 10-Year Follow-Up of Patients With Everolimus-Eluting Versus Bare-Metal Stents After ST-Segment Elevation Myocardial Infarction. J Am Coll Cardiol. 2021 Mar 9;77(9):1165-1178. doi: 10.1016/j.jacc.2020.12.059. PMID 33663733

DOCUMENTS (2):
  • Study Protocol (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT04462315/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT04462315/SAP_001.pdf